CLINICAL TRIAL: NCT04793971
Title: Minimal Invasive Treatment of Achilles Tendinopathy: Focus on Percutaneous Release (Maffulli)
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57392
Record Dates: First submitted 2015-03-23; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Tendinopathy
Keywords: chronic midportion Achilles tendinopathy; percutaneous paratenon release
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- postoperative cases: patients that underwent percutaneous release of the paratenon for chronic midportion Achilles tendinopathy
  Interventions: Procedure: percutaneous paratenon release

INTERVENTIONS:
Procedure: percutaneous paratenon release — percutaneous paratenon release for chronic midportion Achilles tendinopathy

SUMMARY:
To evaluate the outcome of percutaneous paratenon release for chronic midportion Achilles tendinopathy.

DETAILED DESCRIPTION:
Since 2011 the percutaneous procedure took the place of the open release of the paratenon for the surgical treatment for chronic midportion Achilles tendinopathy in the investigators' center. In this study the investigators re-evaluate the patients undergoing percutaneous surgery since then in order to compare the outcome with the excellent results cited in literature. The patients will be contacted and asked to participate completing a VAS-score, a VISA-A score and agreeing with a clinical examination.

Approving by the Ethical Committee of UZLeuven is pending.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent percutaneous paratenon release for chronic midportion Achilles tendinopathy

Exclusion Criteria:

* insertional tendinopathy
* open intervention
* (partial) Achilles tendon rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients that underwent percutaneous paratenon release for chronic midportion Achilles tendinopathy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
VISA-A-score | 3 months
  specific questionnaire about (mal-)function of Achilles tendon

SECONDARY OUTCOMES:
SF-36-score | 3 months
  questionnaire about well-being
VAS-score | 3 months
  questionnaire about pain

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matricali, MD, PhD, Principal Investigator — Foot and ankle surgeon
Locations (1):
- University Hospitals of Leuven, Pellenberg, Vlaams-Brabant, Belgium